CLINICAL TRIAL: NCT02394405
Title: Myocardial and Renal Dysfunction by Oxidative Stress Caused by Cardiac Surgery
Status: Terminated | Type: Observational
Sponsor: Moscow Regional Research and Clinical Institute (MONIKI) (Other Government)
Responsible Party: Principal Investigator, Valery V. Likhvantsev, Professor, senior researcher, Moscow Regional Research and Clinical Institute (MONIKI)
Other Study IDs: OD-CABG-2015
Record Dates: First submitted 2015-02-12; First posted 2015-03-20 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- valve surgery: valve plasty/replacement surgery
- off-pump CABG: off-pump CABG
- CPB-CABG: CABG with CardioPulmonal Bypass

SUMMARY:
Assessment of the severity of oxidative stress caused by the on-pump and off-pump cardiac surgery using mtDNA, nDNA, carbonilated proteins, nitrotyrosine, oxy-LDL, S100b-protein.

ELIGIBILITY:
Inclusion Criteria:

* shedduled CABG

Exclusion Criteria:

* stroke befor surgery
* miocardial infarction 6 monthes befor surgery
* dementia
* liver cirrhosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Assay of mtDNA | from baseline whithin 72 hours

SECONDARY OUTCOMES:
Assay of nDNA | from baseline whithin 72 hours
Assay of carbonilated proteins | from baseline whithin 72 hours
Assay of nitrotyrosine | from baseline whithin 72 hours
Assay of oxy-LDL | from baseline whithin 72 hours
Assay of S100b-protein | from baseline whithin 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow Regional Research and Clinical Institute Moniki n.a. M.F. Vladimirskiy, Moscow, Russia